CLINICAL TRIAL: NCT04968600
Title: Gait Pattern Comparison of Cruciate-retaining and Posterior-stabilized Total Knee Arthroplasties: Gait Analysis With a Smartphone Application
Brief Title: Gait Pattern Comparison of Cruciate-retaining and Posterior-stabilized Arthroplasties
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Deniz CANKAYA, Associate Professor, Gulhane Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021/15
Record Dates: First submitted 2021-07-05; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Knee Osteoarthritis
Keywords: knee arthroplasty; gait analysis; smart-phone
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterior-cruciate-ligament-retaining (CR) (Experimental): Posterior-cruciate-ligament-retaining (CR) technique of total knee arthroplasty
  Interventions: Procedure: total knee arthroplasty
- posterior-cruciate-ligament-stabilized (PS) (Experimental): Posterior-cruciate-ligament-retaining (CR) technique of total knee arthroplasty
  Interventions: Procedure: total knee arthroplasty

INTERVENTIONS:
Procedure: total knee arthroplasty — Posterior-cruciate-ligament is retained in one arm and sacrificed in another arm during total knee arthroplasty

SUMMARY:
In total knee arthroplasty (TKA), the posterior-cruciate ligament-retaining (CR) and posterior-cruciate-ligament stabilized (PS) techniques are widely used depending on the individual preference of the surgeon. Comparative analysis of these two techniques is a major topic of investigation in arthroplasty research. The hypothesis of the present study is that compared with the CR technique, the PS technique is associated with a worse gait pattern. Smart-phone based gait analysis and patient-reported functional outcomes are evaluated in patients undergoing total knee arthroplasty with a CR and a PS technique, at 3, 6, and 12 months postoperatively.

DETAILED DESCRIPTION:
Patients undergoing total knee arthroplasty are randomized to posterior-cruciate ligament-retaining (CR) and posterior-cruciate-ligament stabilized (PS) groups by generating random numbers with Microsoft Excel. The patients are/will be evaluated preoperatively and at 3, 6, and 12 months postoperatively, with knee scores (KSS and KOOS), life quality (SF-12), and smart-phone based gait analysis. All data will be calculated as mean and standard deviation values. The Student's t-test will be used for statistical analysis of the patient data. Statistical calculations will be performed using SPSS vn.22.0 software (IBM SPSS Statistics for Windows, Version 22.0. Armonk, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of unilateral primary knee osteoarthritis
* Age 55 to 85 years
* Must be able to walk without support

Exclusion Criteria:

* Rheumatological joint diseases
* Previous knee surgery
* Neuromuscular diseases
* Bilateral knee osteoarthritis
* Insufficiency of knee collateral ligaments.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
smart-phone based gait analysis | Change from preoperative gait analysis at 3rd month gait analysis
  Gait analysis is made using the Gait Analyzer version 0.9.95.0 (Control One LLC, NM, USA) smartphone application
smart-phone based gait analysis | Change from 3rd month gait analysis at 6th month gait analysis
  Gait analysis is made using the Gait Analyzer version 0.9.95.0 (Control One LLC, NM, USA) smartphone application
smart-phone based gait analysis | Change from 6th month gait analysis at 12th month gait analysis
  Gait analysis is made using the Gait Analyzer version 0.9.95.0 (Control One LLC, NM, USA) smartphone application

SECONDARY OUTCOMES:
Knee functional scores | Change from preoperative Knee Society Scores (KSS) at 3rd month Knee Society Score (KSS)
  Knee Society Score (KSS) (has two different subscale : Knee and Function 100-80: Excellent 79-70:Good 69-60:Fair below 60:Poor )
Knee functional scores | Change from 3rd month Knee Society Scores (KSS) at 6th month Knee Society Score (KSS)
  Knee Society Score (KSS) (has two different subscale : Knee and Function 100-80: Excellent 79-70:Good 69-60:Fair below 60:Poor )
Knee functional scores | Change from 6th month Knee Society Scores (KSS) at 12th month Knee Society Score (KSS)
  Knee Society Score (KSS) (has two different subscale : Knee and Function 100-80: Excellent 79-70:Good 69-60:Fair below 60:Poor )

CONTACTS AND LOCATIONS:
Overall Officials: Deniz CANKAYA, Assoc.Prof., Study Chair — Gulhane Teaching and Research Hospital; Denizhan SIVRI, MD, Principal Investigator — Gulhane Teaching and Research Hospital
Locations (1):
- Gulhane Teaching and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No